CLINICAL TRIAL: NCT04523857
Title: A Phase II Pilot Trial of ABemacicliB or Abemaciclib and HydroxYchloroquine to Target Minimal Residual Disease in Breast Cancer Patients ("ABBY")
Brief Title: ABemacicliB or Abemaciclib and HydroxYchloroquine to Target Minimal Residual Disease in Breast Cancer
Acronym: ABBY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 10119
Record Dates: First submitted 2020-08-06; First posted 2020-08-24 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — abemaciclib; Hydroxychloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- A (Abema) (Experimental): Abemaciclib (150 mg BID)
  Interventions: Drug: Abemaciclib
- B (Abema + HCQ) (Experimental): Abemaciclib (100 mg or 150 mg BID*) + Hydroxychloroquine (600 mg BID)
  *Abemaciclib dose will be determined by safety cohort
  Interventions: Drug: Abemaciclib; Drug: Hydroxychloroquine

INTERVENTIONS:
Drug: Abemaciclib — Oral CDK4/6 inhibitor to target bone marrow disseminated tumor cells (DTCs)
  Other Names: Verzenio
Drug: Hydroxychloroquine — Oral autophagy inhibitor to target bone marrow disseminated tumor cells (DTCs)
  Other Names: Plaquenil
  Arms: B (Abema + HCQ)

SUMMARY:
This is a Phase II randomized, controlled, open label breast cancer clinical trial. 66 patients will be enrolled. The drugs being studied are hydroxychloroquine (Plaquenil) and abemaciclib (also Verzenio). This research study is testing whether using these drugs to target the disseminated tumor cells in bone marrow can reduce their number or eliminate them. Both hydroxychloroquine and abemaciclib are pills that will be taken twice daily. Both are approved by the FDA

ELIGIBILITY:
Inclusion Criteria:

* Histologically-confirmed, primary, invasive breast cancer diagnosed within 5 years of entry into the companion DTC screening protocol UPCC 28115
* Qualifying risk status, at diagnosis utilizing receptor testing by ASCO/CAP guidelines, meting at least one of the following:

  (i) Histologically positive axillary lymph nodes, regardless of receptors (ii) Primary tumor that is ER/PR/Her2 negative: estrogen receptor (ER) < 10%, progesterone receptor (PR) < 10% and negative for Her2-overexpression by ASCO-CAP guidelines, regardless of lymph nodes status (iii) Primary tumor that is ER+/Her2 negative/Lymph node negative with Breast Cancer Recurrence Score of >/= 25 per the Genomic Health Oncotype DX breast cancer test and/or high risk MammaPrint (iv) Evidence of residual disease in the breast on pathologic assessment after neoadjuvant chemotherapy
* Patients must have completed all primary therapy (definitive surgery, (neo)adjuvant chemotherapy adjuvant radiation and/or Her2-directed therapy) for the index malignancy at least 4 weeks prior to study entry. Prior treatment-related toxicity must be resolved or improving to Grade 1 with the exception of alopecia, Grade 2 endocrine disorders (e.g. adrenal insufficiency or thyroid disorders from prior immunotherapy) controlled on stable replacement therapy for > 1 year, and up to Grade 3 peripheral neuropathy, prior to study enrollment. Concurrent receipt of adjuvant endocrine and bone modifying agents is allowed per standard of care guidelines. Tamoxifen is not allowed due to drug-drug interactions with HCQ.
* Bone marrow aspirate obtained via research trial UPCC 28115 after completion of therapy (except endocrine therapy) demonstrates detectable DTCs (via IHC)
* No evidence of recurrent local or distant breast cancer by physical examination, blood tests (CBC, LFTs, Alk Phos), or imaging. Assessment for overt metastatic disease by radiologic testing per institutional guidelines (CT Chest, Abdomen and Pelvis, bone scan, MRI and/or PET/CT) will only be done in patients with DTCs detected on bone marrow aspirate who are being screened for this trial.
* Age >/= 18 years
* ECOG performance status =/< 2
* Ability to swallow oral medications
* No contraindications to the study medications or uncontrolled medical illness.
* Adequate bone marrow function as shown by: ANC >/= 1.5 x 10^9/L, Platelets >/= 100 x 10^9/L, Hb >9 g/dL
* Adequate liver function as shown by: Serum bilirubin </= 1.5 x ULN, ALT and AST </= 3.0 x ULN, and INR </=1.5
* Adequate renal function: serum creatinine </= 1.5 x ULN
* Adequate muscle function: creatinine phosphokinase (CPK) </= 2.5 x ULN
* Anticoagulation is allowed if target INR =/< 1.5 on a stable dose of warfarin or on a stable dose of anticoagulant for >2 weeks at time of randomization
* Ability to provide informed consent

Exclusion Criteria

* Concurrent enrollment on another investigational therapy
* Patient has received an experimental treatment in a clinical trial within the last 30 days or 5 half-lives, whichever is longer, prior to randomization (or treatment assignment), or is currently enrolled in any other type of medical research (for example: medical device) judged by the sponsor not to be scientifically or medically compatible with this study.
* Prior treatment with a CDK 4/6 inhibitor
* Known hypersensitivity to hydroxychloroquine or any of its derivatives
* Prior hydroxychloroquine exposure for a duration of > 1 month since the completion of the patient's primary therapy (definitive surgery, (neo)adjuvant chemotherapy, adjuvant radiation, and/or Her2-directed therapy) for the index malignancy.
* Patients with hormone-receptor positive breast cancer may not be receiving tamoxifen due to drug-drug interactions with hydroxychloroquine
* Patients who have initiated bone modifying agents within 3 months prior to the start of study treatment
* Patients who have had major surgery within 14 days prior to randomization (or treatment assignment)
* Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study
* Female patients who are pregnant or breast feeding, or adults of reproductive potential who are not using effective birth control methods.
* Women of childbearing potential must have a negative serum pregnancy test within 7 days prior to the first dose of Abema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events during cycle 1 of the safety cohort (safety of combination HCQ + Abema) | Toxicity is assessed over the first cycle (4 weeks) of treatment
  Rate of protocol defined "severe toxicity" during cycle 1 (4 weeks) of combination HCQ 600mg BID and Abema (at 100 mg and 150 mg BID) in a safety cohort of 6 patients at each dose of Abema
Change in bone marrow DTC number evaluated by DTC-IHC assay after 6 cycles of therapy compared to baseline (Efficacy of Abema +/- HCQ in eliminating bone marrow DTCs) | 6 cycles (approximately 6 months)
  Frequency of "clearance" of bone marrow DTCs by arm after 6 cycles of study treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Amy Clark, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States